CLINICAL TRIAL: NCT01803516
Title: Quality of Life Assessment in Breast Cancer Patients With Radiation-Induced Telangiectasias Treated With the Pulsed Dye Laser
Brief Title: QOL Assessment in Breast Cancer Patients With Radiation-Induced Telangiectasias Treated With the Pulsed Dye Laser
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 13-013
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer; Radiation-Induced Telangiectasias
Keywords: Quality of Life; Assessments; Radiation; Telangiectasias; 13-013
MeSH Terms: conditions — Breast Neoplasms; Telangiectasis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Breast cancer survivors with radiation-induced Telangiectasias: A quality of life assessment will also be completed by the patient using the Skindex-16 and a subscale of the BREAST-Q Breast Conserving Module questionnaire.
  Interventions: Behavioral: questionnaires

INTERVENTIONS:
Behavioral: questionnaires — This study will be offered to patients who, at the time of consultation are identified as having had adjuvant breast radiation treatment following surgical treatment for breast cancer and developed radiation-induced telangiectasias. The Skindex-16 and BREAST-Q questionnaires will be used to evaluate the quality of life of The study participants. For each instrument, for each evaluation time point, QOL scores will be summed and transformed into a scale from 0-100. Descriptive statistics will be used to describe the QOL of the study participants.

SUMMARY:
The purpose of this study is to see how the look of telangiectasias (small dilated blood vessels) on radiated breast skin when altered by the pulsed dye laser affects a patient's overall well being.

Patients will have a set of treatments with a pulsed dye laser. This is a laser that targets red blood vessels and delivers heat causing the telangiectasias to become smaller and less visible. The laser has been used safely to treat telangiectasias on the skin of patients who received radiation for breast cancer.

Patients in the study will be asked to complete a questionnaire asking how they feel about the telangiectasias, their radiated skin and its effect on their daily lives. The questionnaire will be given at every visit. The improvement in the look of patients' radiated skin will also be compared to answers to the questionnaire. We hope the study will improve our understanding of how patients feel about the long term effects of radiation on their skin.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced breast cancer patients treated with surgery and adjuvant radiation
* Telangiectasias in the radiation field of the treated breast
* Patients 18 years or older

Exclusion Criteria:

* Non English speaking
* Current oral steroid use or receiving daily therapeutic anticoagulation (e.g. Coumadin, Lovenox)
* Breast/s reconstructed with implant in the area of previous radiation
* Pregnancy or lactation
* Previous laser treatment of telangiectasias
* Presence of a sun tan in the area
* Fitzpatrick skin types V, VI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Dermatology Division and/or Radiation Oncology, Plastic and Reconstructive Surgery Department(s) and the Breast Cancer Survivorship Program will be identified by the Nurse Practitioners of the survivorship program or by clinicians in these departments for the study.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2013-02; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
evaluate quality-of-life (QoL) | 2 years
  in breast cancer survivors with chronic radiation-induced telangiectasias who are undergoing pulsed dye laser treatment. To assess quality of life in relation to the radiation-induced telangiectasias, two pre-existing validated scales will be utilized. The Skindex-16 and BREAST-Q are scales that have been validated to assess quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Lee, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/